CLINICAL TRIAL: NCT03067870
Title: Transplantation of Autologous Purified Bone Marrow Derived Specific Populations of Stem Cells and Mesenchymal Stem Cells in Patients With Rheumatoid Arthritis
Brief Title: Transplantation of Autologous Bone Marrow Derived Stem Cells in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stem Cells Arabia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA-RA1
Record Dates: First submitted 2017-02-25; First posted 2017-03-01 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: RheumatoId Arthritis; Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Stem cells; Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cells (Experimental): Autologous bone marrow-derived stem cell transplantation.
  Interventions: Biological: Stem Cell Transplantation

INTERVENTIONS:
Biological: Stem Cell Transplantation — * Intravenous administration of autologous bone marrow derived stem cells for immunomodulation.
  * Transplantation of autologous bone marrow derived stem cells in joints.

SUMMARY:
Rheumatoid arthritis is a chronic systemic disease, which is characterized by chronic inflammation in the synovial tissue. Rheumatoid arthritis ultimately results in the destruction of cartilage, bone and ligaments and joint deformity. The underlying hypothesis is that autologous bone marrow-derived mesenchymal and specific populations of stem cells has anti-inflammatory and regenerative effects and thus potentially alleviates the progression of rheumatoid arthritis. The study is to explore the safety and efficacy of BM-SC transplantation in treatment of rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic autoimmune disorder that primarily affects joints. It typically results in swollen and painful joints. Pain and stiffness often worsen after rest. Most frequently, the wrist and hands are involved, with the same joints typically involved on both sides of the body. RA affects between 0.5-1% of adults in the developed world with between 5-50 per 100,000 people newly developing the disease each year. Onset is most frequent during middle age and women are affected 2.5 times as frequently as men. The goal of treatment is to reduce pain, decrease inflammation, and improve a person's overall functioning and quality of life.

Herein, the investigators study the safety and efficacy of the immunomodulatory effects of bone marrow-derived stem cells administered intravenously and the regenerative and repair potential of bone marrow-derived stem cells transplanted into the joints of patients with RA.

ELIGIBILITY:
Inclusion Criteria:

* 17-75 years old
* The presence of osteoarthritis based on MRI and American Rheumatism Association criteria since 6 months before treatment.

Exclusion Criteria:

* Subjects with addition major health condition/disease diagnoses
* Subjects that are pregnant or breastfeeding

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Pain Reduction measured by VAS scaling | 1 month
  measured by VAS scaling

SECONDARY OUTCOMES:
Evaluation of the Physical Activity measure by WOMAC scoring | 1 month
Evaluation the resurfacing of articular cartilage by MRI | 6 months

IPD SHARING:
Plan to Share IPD: Undecided